CLINICAL TRIAL: NCT05024266
Title: Tislelizumab Combined With Albumin Paclitaxel + Carboplatin as Neoadjuvant Therapy for Patients With Stage IIIA-IIIB (N2) Lung Squamous Cell Carcinoma: A Single-arm, Single-center, Exploratory Phase II Clinical Study
Brief Title: Tislelizumab Combined With Chemotherapy as Neoadjuvant Therapy for Stage IIIA-IIIB (N2) Lung Squamous Cell Carcinoma
Acronym: TACT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210011C-R1
Record Dates: First submitted 2021-08-10; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Lung Squamous Cell Carcinoma; Neoadjuvant Therapy; Immunotherapy
Keywords: Lung Squamous Cell Carcinoma; neoadjuvant therapy; immunotherapy
MeSH Terms: interventions — tislelizumab; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab + Albumin Paclitaxel + Carboplatin (Experimental): Tislelizumab 200mg d1, Albumin Paclitaxel 260mg/m2 d1, Carboplatin AUC5 d1, Q3W
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Participants received 2 cycles Tislelizumab 200mg d1 + Albumin Paclitaxel 260mg/m2 d1 + Carboplatin AUC5 d1 every 3 weeks, and then were evaluated for surgery.
  Other Names: Albumin Paclitaxel; Carboplatin

SUMMARY:
Tislelizumab combined with chemotherapy has shown good efficacy and safety in clinical studies of lung adenocarcinoma (RATIONALE 304) and lung squamous cell carcinoma (RATIONALE 307), thus has been approved as the first-line therapy for advanced non-small cell lung cancer (NSCLC) in China. However, there is no data in the field of neoadjuvant therapy for NSCLC. This single-arm, single-center phase II clinical study is designed to evaluate the efficacy, safety and major pathological response (MPR) of Tislelizumab combined with chemotherapy as neoadjuvant therapy in patients with stage IIIA-IIIB (N2) lung squamous cell carcinoma. Biomarkers correlated with efficacy outcomes will also be explored.

DETAILED DESCRIPTION:
Tislelizumab combined with chemotherapy has shown good efficacy and safety in clinical studies of lung adenocarcinoma (RATIONALE 304) and lung squamous cell carcinoma (RATIONALE 307), thus has been approved as the first-line therapy for advanced non-small cell lung cancer (NSCLC) in China. However, there is no data in the field of neoadjuvant therapy for NSCLC. This single-arm, single-center phase II clinical study intends to enroll about 30 patients with potentially operable lung squamous cell carcinoma with clinical stages IIIA-IIIB (N2). Participants will intravenously receive tislelizumab (BeiGene, 200mg d1) + albumin paclitaxel 260mg/m2 d1 + carboplatin AUC 5 d1, Q3W, Imaging evaluation is performed after 2 cycles of medication, and the feasibility of surgery is discussed in multiple disciplines. If the evaluation is operable, the lesion will be surgically removed 22-40 days after the last treatment. If it is assessed to be reduced but still inoperable, the original plan will be continued for another cycle. Imaging examinations, tissue NGS (whole-exome sequencing), gene expression profiling (GEP), and PD-L1 expression will be performed at baseline, preoperative and postoperative respectively.

ELIGIBILITY:
Inclusion Criteria:

1. The age is ≥18 years old and <75 years old.
2. Eastern Cooperative Oncology Group (ECOG) physical status is 0 or 1.
3. Untreated and histologically confirmed squamous cell lung carcinoma.
4. Potentially operable stage IIIA-IIIB (N2) squamous cell lung carcinoma on enrollment (as defined by the American Joint Committee on Cancer 8th Edition).
5. Sufficient pre-treatment tumor tissue samples/peripheral blood samples for biomarker analysis.
6. Sufficient organ functions, including: Haematological status: absolute neutrophil count(ANC) ≥1.5×10^9 /L, platelet count(PLT) ≥100×10^9 /L, hemoglobin(HB) ≥90 g/L; Liver function: alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤2.5 x upper limit of normal range (ULN), total bilirubin (TBIL)≤1.5 x upper limit of normal range (ULN); Kidney function: Creatinine(Cr)≤1.5 x upper limit of normal range(ULN) or Creatinine clearance ≥45 ml/min (calculated according to Cockcroft-Gault equation)

Exclusion Criteria:

1. Participants with known EGFR, ALK or ROS1 sensitive mutations.
2. Participants with autoimmune diseases, tuberculosis, active hepatitis or HIV.
3. Participants who are not expected to tolerate surgery, such as patients with cardiopulmonary insufficiency, etc.
4. A history of other malignant tumors in the past 5 years, except for cured cervical carcinoma in situ, cured basal cell carcinoma of the skin and superficial bladder cancer [Ta, Tis & T1].
5. Participants who have used PD-1/PD-L1 and other immunotherapy drugs before.
6. Women of childbearing age as the exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | 2-4 weeks after resection
  Major Pathological Response (MPR) is evaluated after resection by pathologists, which is defined as a metric of ≤10% residual tumor tissue after neoadjuvant therapy.
Incidence of Treatment-Emergent Adverse Events | Through the trial
  Adverse events are evaluated by investigators according to CTCAE 5.0.

SECONDARY OUTCOMES:
Rate of radical resection (R0) | 4 weeks after resection
  The rate of radical resection (R0) is evaluated by the investigator, which is the number of participants who can undergo R0 resection after the evaluation criteria established by the MDT team divided by the total number of enrolled groups.
Overall Response Rate (ORR) | 4 weeks after resection
  The overall response rate is evaluated by the investigator, which is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set (e.g. efficacy evaluable population)
Disease-free survival (DFS) | 1 year and 2 years after resection
  Disease-free survival (DFS) is evaluated by the investigator, which is the percentage of individuals in the treatment group who are likely to be free of the signs and symptoms of a disease after a specified duration of time.
Overall survival (OS) | Through the trial
  Overall survival (OS) evaluated by the investigator, which is the percentage of people in a group who are alive after a length of time.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shan J, Liu Z, Chen S, Du C, Li B, Ruan L, Kong M, Wang L, Du M, Shi S, Qiao G, Tian T, Tu Z. Optimizing perioperative treatment for potentially resectable stage III squamous cell lung carcinoma: promising results of a condensed four-cycle regimen with tislelizumaband chemotherapy. BMC Med. 2024 Jun 10;22(1):234. doi: 10.1186/s12916-024-03462-4. PMID 38853265